CLINICAL TRIAL: NCT04296864
Title: A Multi-Center, Double-Masked, Randomized, Placebo-Controlled, Parallel-Group Study Evaluating the Efficacy, Safety, and Tolerability of Dupilumab in Patients With Atopic Keratoconjunctivitis (AKC)
Brief Title: Evaluation of Dupilumab in Patients With Atopic Keratoconjunctivitis (AKC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andover Eye Associates (Industry)
Collaborators: Statistics & Data Corporation (Industry); Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-290-0002
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Atopic Keratoconjunctivitis
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double-masked study in which both participants and investigators will be masked to study treatment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo of Dupilumab
  Interventions: Drug: Dupilumab
- Dupilumab (Experimental): one loading dose of Dupilumab 600 mg followed by Dupilumab 300 mg weekly for a total of 16 weeks
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — monoclonal antibody
  Other Names: Dupixent

SUMMARY:
This is a multi-center, double-masked, randomized, placebo-controlled, parallel-group, efficacy, safety, and tolerability study evaluating the efficacy of Dupilumab in the treatment of signs and symptoms of atopic keratoconjunctivitis (AKC).

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age at Visit 1 of either gender and any race or ethnicity;
* provide written informed consent and sign the HIPAA form;
* be willing and able to follow all instructions and attend all study visits;
* if on an active therapy for AKC prior to Visit 1, such treatment must have been maintained stably for at least 2 weeks for topical corticosteroids, topical and oral antihistamines, topical mast cell stabilizers, and topical tacrolimus and at least 3 months for topical and oral cyclosporine, and systemic corticosteroids. Such therapy must remain current throughout duration of study;
* have a history of AKC or atopic dermatitis with a diagnosis of AKC at Visit 1 (by meeting inclusion 7 and 8);
* be able to self-administer or receive subcutaneous injections satisfactorily or have a caregiver at home routinely available for this purpose. If unable to administer at home, patients must be willing to come in to office to receive injections that do not coincide with a visit;
* present signs of active disease, defined as one or more of the following in at least one eye at Visit 2 (baseline):

  1. >/=2 score in conjunctival redness AND
  2. >/=2 score in at least one of the following lid disease signs: i. lid margin redness ii. lid excoriation
* present symptoms of active disease, defined as having both of the following in at least one eye at Visit 2 (baseline):

  1. >/=2.5 score in ocular itching AND
  2. >/=2 score for ocular discomfort;
* (for females capable of becoming pregnant) agree to have urine pregnancy testing performed at screening (must be negative) and at exit visit; must not be lactating; and must agree to use at least one medically acceptable form of birth control throughout the study duration and for at least 14 days prior to the first dose of investigational product (Visit 2) and for 1 month after the last dose of investigational product. Note: Women considered capable of becoming pregnant include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy);
* have a calculated visual acuity of 0.7 logarithm of the minimum angle of resolution (logMAR) or better in at least one eye (Snellen equivalent of 20/100) and 1.0 logMAR (or count fingers) or better in the fellow eye (Snellen equivalent of 20/200) as measured using an Early Treatment for Diabetic Retinopathy Study (ETDRS) chart.

Exclusion Criteria:

* have known contraindications or sensitivity to the use of any of the study drug(s) or their components, or any other medications required by the protocol;
* wear contact lenses for at least 48 hours prior to and during the study trial period;
* have a corneal ulcer in either eye;
* have a presence or history of ocular herpes or varicella-zoster infections in either eye;
* have uncontrolled ocular hypertension or glaucoma in either eye;
* have prior (within 30 days of beginning investigational product) or anticipated concurrent use of an investigational product or device during the study period;
* have an ocular or systemic condition or a situation which, in the investigator's opinion, may put the patient at increased risk, confound study data, or interfere significantly with the patient's study participation;
* manifest in either eye symblepharon, significant conjunctival scarring, and/or fornix shortening;
* have planned surgery (ocular or systemic) during the trial period or within 30 days after the study period;
* have an abnormal blood pressure (defined as ≤ 90 or ≥ 160 (systolic) measured in mmHg or ≤ 60 or ≥ 100 (diastolic) measured in mmHg) at Visit
* be a female who is currently pregnant, planning a pregnancy, or lactating;
* have any previous exposure to dupilumab (unless discontinuation of exposure was due to a non-medical reason);
* have treatment with a live (attenuated) vaccine during the study;
* have an untreated parasitic (helminth) infection prior to Visit 2 and during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of treatment responders | Baseline to Week 16
  • Determination of the percentage of treatment responders as defined as meeting one or more of the below at the end of the 16-week treatment period (Visit 7) as compared to Visit 2 (baseline):
  * ≥ 1 grade improvement in lid margin redness (0-3 scale, NOT allowing half unit increments)
  * ≥ 1 grade improvement in lid excoriation (0-3 scale, NOT allowing half unit increments)
  * ≥ 1 grade improvement in lid thickening/lichenification (0-3 scale, NOT allowing half unit increments)
  * ≥ 1 grade improvement in changes in mucocutaneous junction (0-3 scale, NOT allowing half unit increments)
  * ≥ 4 grade improvement in a composite symptom score (the sum of scores for ocular itching, tearing/watery eyes, ocular discomfort, photophobia, and nonpurulent mucous discharge)
  * >2 grade improvement in an individual symptom from Visit 2 (baseline)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Premiere Practice Management, LLC, Los Angeles, California
  - Colorado Eye Consultants/Corneal Consultants of Colorado, Littleton, Colorado
  - Encore Medical Research, LLC, Hollywood, Florida
  - Kannar Eye Care, Pittsburg, Kansas
  - Andover Eye Associates, Andover, Massachusetts
  - University of Michigan- Kellogg Eye Center, Ann Arbor, Michigan
  - Silverstein Eye Centers, Kansas City, Missouri
  - Mercy Clinic Eye Specialists, Springfield, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - St. Louis Eye Institute, Town and Country, Missouri
  - Northwell Health Physician Partners Ophthalmology at Great Neck, Great Neck, New York
  - Gerald W. Zaidman, MD, Hawthorne, New York
  - NC Eye Associates, Apex, North Carolina
  - Vita Eye Clinic, Shelby, North Carolina
  - Tracie Malsom, Fargo, North Dakota
  - Vantage EyeCare, LLC., Bala-Cynwyd, Pennsylvania
  - Blink Research Center, Memphis, Tennessee
  - Advancing Vision Research, LLC, Smyrna, Tennessee
  - Eye Associates of Central Texas, Round Rock, Texas
  - Periman Eye Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No